CLINICAL TRIAL: NCT04629807
Title: The Anterior Gen Plus Study
Brief Title: Anterior Gen Plus Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS-OS-1901
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Spine Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Demineralized Bone Matrix (DBM) (Active Comparator): All enrolled subjects will undergo primary, contiguous 2-level ALIF without supplemental fixation. Study Implant (one-level) implanted with Demineralized Bone Matrix (DBM).
  Interventions: Procedure: Anterior Lumbar Interbody Fusion (ALIF)
- Cellular Bone Matrix (CBM) (Active Comparator): All enrolled subjects will undergo primary, contiguous 2-level ALIF without supplemental fixation. Control Implant (one-level) implanted with Cellular Bone Matrix (CBM).
  Interventions: Procedure: Anterior Lumbar Interbody Fusion (ALIF)

INTERVENTIONS:
Procedure: Anterior Lumbar Interbody Fusion (ALIF) — Intra-Operative Anterior Lumbar Interbody Fusion (ALIF)

SUMMARY:
A clinical study evaluating patients treated with the Demineralized Bone Matrix (DBM) as compared to a Cellular Bone Matrix (CBM) in anterior lumbar interbody fusion.

DETAILED DESCRIPTION:
A prospective, single-center, clinical study evaluating patients undergoing primary, contiguous 2-level ALIF without supplemental fixation treated with Demineralized Bone Matrix (DBM) as compared to a Cellular Bone Matrix (CBM).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Requires anterior lumbar interbody (ALIF) fusion
* Are physically and mentally able and willing to return for the scheduled follow up visits, follow post-operative instructions
* Willing and able to sign study specific Informed Consent Form

Exclusion Criteria:

* Signs of acute infection
* Active malignancy and/or current chemotherapy
* Prior fusion at operative or adjacent level
* Institutionalized or a prisoner
* Documented history of alcohol or drug abuse
* Undergoing a worker's compensation case
* Pregnancy
* Participation in another research study involving another implant or drug that may affect the outcomes of this clinical study
* Any other condition that the Investigator determines is unacceptable for enrollment into this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of fusion for the DBM versus CBM cohorts | 12 months
  Proportion of levels exhibiting fusion for the DBM cohort versus the CBM cohort

SECONDARY OUTCOMES:
Serious Adverse Events (SAEs) | 24 Months
  SAEs at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Muwaffak Abdulhak, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No